CLINICAL TRIAL: NCT06951711
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of KarXT for the Treatment of Manic Episodes in Bipolar-I Disorder (BALSAM-2)
Brief Title: A Study to Evaluate the Efficacy and Safety of KarXT for the Treatment of Manic Episodes in Bipolar-I Disorder (BALSAM-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN012-0037; 2024-520195-94 (Other: EU CTR); U1111-1316-7466 (Other: WHO)
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Disorder Type I With Mania or Mania With Mixed Features
Keywords: Bipolar-I disorder; Mania; Bipolar-I disorder with Mania
MeSH Terms: conditions — Mania | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental): Flexible dosing
  Interventions: Drug: KarXT
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510; Xanomeline and trospium chloride
  Arms: KarXT
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled, multicenter, inpatient study in participants with bipolar disorder experiencing an acute episode of mania or mania with mixed features.

The primary objective of the study is to evaluate the efficacy of KarXT compared to placebo in treating symptoms of mania during a 3-week inpatient period. The duration of the study including screening, the double-blind inpatient treatment period and safety-follow-up is no more than seven weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a primary diagnosis of Bipolar-I disorder established by a comprehensive psychiatric evaluation.
* Participants must be experiencing an acute episode or relapse of mania or mania with mixed features (≤ 3 weeks).
* Participants must require hospitalization for the acute exacerbation or relapse of mania.
* Participants must have all psychotropic medications washed out in no more than 14 days prior to the first dose of the study drug.
* Participants must have a Young Mania Rating Scale (YMRS) score of ≥ 20 at Screening and at Baseline.
* Participants must have a Clinical Global Impressions-Bipolar (CGI-BP) ≥ 4 at Screening and at Baseline.

Exclusion Criteria:

* Participants must not have any primary Diagnostic and Statistical Manual of Mental Disorders (5th Edition, Text Revision) (DSM-5-TR) disorder, other than BP-I with mania or mania with mixed features within 12 months before screening, including BP-I with depression (for previous 3 months only), BP-II disorder, borderline personality disorder, major depressive disorder, and primary psychotic disorder, with the exception of mild anxiety disorders.
* Participants must not have a primary diagnosis of BP-I with rapid cycling (≥ 4 distinct mood episodes in one year).
* Participants must not have a DSM-5-TR diagnosis of moderate to severe substance use disorder (except tobacco use disorder) within the 12 months before screening, or current use as determined by urine toxicology screen or alcohol test.
* Participants must not be at risk for suicidal behavior at screening or the baseline visit as determined by the Investigator's clinical assessment and the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Participants must not have cirrhosis, liver cancer, clinically significant liver disease based on the liver function test results.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Young Mania Rating Scale (YMRS) score | At week 3
  The YMRS comprised of 11 items that assess the severity of manic symptoms. All items are given a severity rating, with 4 items graded from 0 to 8 (irritability, speech, thought content, and disruptive/aggressive behavior), and the remaining 7 items are graded from 0 to 4 points. The highest score obtainable on the YMRS is 60 and the higher the number the greater the number of symptoms and/or the greater their severity.

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impressions-Bipolar (CGI-BP) | At week 3
  The CGI-BP is designed to assess the severity, improvement, and efficacy of treatment in individuals with bipolar disorder. Only section I, illness severity, will be used, which includes three components: mania, depression, and overall bipolar illness. The ratings are on a 7-point scale (1 = normal, not ill; 2 = minimally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = very severely ill).
Occurrence of response based on ≥ 50% decrease from baseline in YMRS score or total score | At week 3
Occurrence of response based on change from baseline ≥ 1 in CGI-BP | At week 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (64):
- United States (27):
  - Pillar Clinical Research- Little Rock, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Proscience Research Group, Culver City, California
  - Clinical Innovations, Inc. dba CITrials, Riverside, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Local Institution - 0036, Hialeah Gardens, Florida
  - Behavioral Clinical Research, Hollywood, Florida
  - LCC Medical Research Institute, Miami, Florida
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida
  - Health Synergy Clinical Research, Stuart, Florida
  - Local Institution - 0019, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Local Institution - 0020, Chicago, Illinois
  - CBH Health, Gaithersburg, Maryland
  - Local Institution - 0017, Flowood, Mississippi
  - Arch Clinical Trials, St Louis, Missouri
  - Local Institution - 0076, North Las Vegas, Nevada
  - Hassman Research Institute Marlton Site, Marlton, New Jersey
  - Local Institution - 0031, Marlton, New Jersey
  - Local Institution - 0075, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - InSite Clinical Research, DeSoto, Texas
  - Local Institution - 0028, Houston, Texas
  - Pillar Clinical Research - Richardson, Richardson, Texas
- Croatia (5):
  - Local Institution - 0009, Zagreb, City of Zagreb
  - Local Institution - 0008, Zagreb
  - Local Institution - 0010, Zagreb
  - Local Institution - 0063, Zagreb
  - Local Institution - 0078, Zagreb
- India (7):
  - Local Institution - 0065, Vadodara, Gujarat
  - Local Institution - 0082, Belagavi, Karnataka
  - Local Institution - 0053, Kozhikode, Kerala
  - Local Institution - 0051, Ludhiana, Punjab
  - Local Institution - 0052, Hyderabad, Telangana
  - Local Institution - 0055, Hyderabad, Telangana
  - Local Institution - 0054, Kolkata, West Bengal
- Israel (6):
  - Shalvata Mental Health Center, Hod HaSharon, Central District
  - Local Institution - 0046, Ness Ziona, Central District
  - Local Institution - 0058, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Be'er Sheva Mental Health Center, Beersheba, Southern District
  - Kfar Shaul Mental Health Center, Jerusalem
- Italy (5):
  - Local Institution - 0001, Milan, Lombardy
  - Local Institution - 0056, Pisa, Tuscany
  - Local Institution - 0007, Siena, Tuscany
  - Local Institution - 0041, Ancona
  - Local Institution - 0040, Genova
- Romania (5):
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital, Bucharest, București
  - Centrul de Evaluare și Tratament a Toxicodependenței pentru Tineri Sf.Stelian, Bucharest
  - Local Institution - 0057, Bucharest
  - Local Institution - 0047, Iași
  - Local Institution - 0061, Sanpetru /Brasov
- Slovakia (3):
  - Local Institution - 0071, Košice, Košice Region
  - Local Institution - 0073, Košice, Košice Region
  - Local Institution - 0072, Vranov nad Topľou, Presov
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Osi Bilbao-Basurto, Bilbao, Basque Country
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
- Sweden (3):
  - Nacka Local Hospital, Nacka, Stockholms Län [se-01]
  - Local Institution - 0067, Uppsala, Uppsala Län [se-03]
  - Local Institution - 0070, Gothenburg, Västra Götalands Län [se-14]

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06951711.html